CLINICAL TRIAL: NCT04307875
Title: Hypertension and Diabetes Mellitus Assessment in the Rohingya Refugee Population and in the Host Communities in Bangladesh
Brief Title: Hypertension and Diabetes Assessment in the Rohingya Refugee Population and in the Host Communities in Bangladesh
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Heidelberg University (Other); Gono Bishwabidyalay (Unknown); Gonoshasthaya Kendra (Unknown)
Responsible Party: Principal Investigator, Dr. Alexander Supady, Principal Investigator, Attending Physician, University Hospital Freiburg
Other Study IDs: coxs_2020
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hypertension; Diabetes Mellitus; Post Traumatic Stress Disorder; Depressive Symptoms
Keywords: Rohingya refugees; Bangladesh; refugee camp
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Stress Disorders, Post-Traumatic; Depression | interventions — Blood Pressure Determination; Psychometrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rohingya refugee camp population: A sample of 1500 randomly selected individuals aged 18 years and above living in the Rohingya refugee camp 1E.
  Interventions: Diagnostic Test: Blood pressure measurement (sphygmomanometer); Diagnostic Test: Blood glucose measurement; Other: psychometric tests
- Shamlapur refugee hosting community population: A sample of 1500 randomly selected individuals aged 18 years and above living in the refugee hosting community Shamlapur neighbouring the Rohingya refugee camps.
  Interventions: Diagnostic Test: Blood pressure measurement (sphygmomanometer); Diagnostic Test: Blood glucose measurement; Other: psychometric tests

INTERVENTIONS:
Diagnostic Test: Blood pressure measurement (sphygmomanometer) — measuring blood pressure with standard sphygmomanometer
Diagnostic Test: Blood glucose measurement — measuring blood glucose using standard measurement devices
Other: psychometric tests — WHODAS 2.0, PHQ-9, CAPS-5

SUMMARY:
Due to a massive outbreak of violence against the Rohingya minority residing in the Rakhine State of Myanmar in late 2017, several hundred thousand Rohingya fled the country and sought a shelter in Bangladesh. Currently, in the refugee settlement areas east of the city of Cox's Bazar, close to 1 million Rohingya refugees live in refugee camps close to the municipalities of Ukhia and Shamlapur.

According to previous examinations, there is a serious burden of non-communicable diseases in Bangladesh. But little is known about the health status and the epidemiology of non-communicable diseases in the Rohingya refugee population in Bangladesh. Most importantly, scientific evidence on non-communicable disease in humanitarian emergencies is rather limited.

The aim of this study is to close this gap and to systematically assess the burden of hypertension and diabetes within the Rohingya refugee population in refugee camps in Bangladesh and in the host community in the Chittagong province. This assessment will help to design and to introduce community-based intervention strategies aiming to improve the population health status and reduce the disease burden.

DETAILED DESCRIPTION:
Cardiovascular diseases are the predominant cause of death globally and in most low- and middle-income countries (LMICs). More than 70% of all global deaths are due to non-communicable diseases, almost half of them are caused by cardiovascular diseases. Diabetes mellitus as a major cardiovascular risk factor accounts for more than 1.5 million global deaths annually (almost 3% of all global deaths). In Bangladesh, according to WHO estimates, 30% of all deaths are due to cardiovascular diseases and 3% are due to diabetes. A recent study on more than 12,338 respondents revealed a 30.1% prevalence of hypertension and a 4.9% prevalence of diabetes among adults aged 35 years and above in Bangladesh.

Due to a massive outbreak of violence against people of the Rohingya minority in the Rakhine state of Myanmar in late 2017 several hundred thousand Rohingya fled the country and sought a refuge in the Chittagong province in south-eastern Bangladesh. These seemingly organized and coordinated attacks have been preceded by massive discrimination and recurrent violence against the Rohingya minority for many decades. Presently, close to 1 million Rohingya refugees settle in the refugee camps in the Chittagong province close to the municipalities of Ukhia and Shamlapur.

Scientific evidence on care of non-communicable diseases (NCDs) in humanitarian emergencies is very limited. A recent systematic review identified only five scientific studies, published between 1980 and 2014 on non-communicable diseases in humanitarian crises. Although many humanitarian organizations from Bangladesh and from abroad organize and support the provision of health services within the refugee camps, systematic evidence on the health status of the Rohingya refugee population is scarce - this is particularly true for chronic and non-communicable diseases.

As in the host community in Bangladesh, there will be a relevant burden of NCDs within the Rohingya refugee population. Furthermore, since the Rohingya have been discriminated for many years and access to health services was restricted for them, many of the diseased will be undiagnosed and untreated and a relevant number of individuals will suffer from long-term complications of untreated disease.

Chittagong province is one of the poorest regions in Bangladesh. Access to primary health services in Bangladesh is limited for many people due to various barriers, affordability being a major reason. A recent observation conducted by Gonoshasthaya Kendra, a project partner in the here presented study, revealed that the distance between place of residence and the nearest health facility and transportation costs are a major obstacle for people in Shamlapur to seek medical care. Data from previous nationwide epidemiologic studies do not sufficiently consider socioeconomic gradients within the Bangladesh population and therefore do not provide substantial information on hypertension and diabetes disease burden in the Rohingya refugee population and the host communities around the refugee camps.

The aim of this study is to systematically assess the burden of hypertension and diabetes mellitus within the Rohingya refugee population in the refugee camps in Bangladesh and in the host community in Chittagong province. This basic epidemiological information is essential for the planning, resource allocation and management of prevention and treatment strategies and programs for the respective populations. Considering the increasing relevance and burden of non-communicable and cardiovascular diseases particularly in low- and middle-income countries, a solid epidemiological data base is a mandatory prerequisite to address this global public health challenge. Therefore, this assessment will help to design and to introduce community-based intervention strategies aiming to improve the population health status and reduce the disease burden.

ELIGIBILITY:
Inclusion Criteria:

* Residing in one of the selected households (Camp 1E or Shamlapur municipality)
* Age ≥18 years

Exclusion Criteria:

* Inability to provide written informed consent
* Participant's unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be a random household sample from Camp 1E at the Cox's Bazar refugee camp area in Bangladesh and a random household sample from the Bangladesh host community in Shamlapur. Camp 1E is located on the northern end of the Cox's Bazar refugee camp area near Ukhia in south-eastern Bangladesh. Shamlapur is a village on the shores of the golf of Bengal, located about 25 kilometers south of Camp 1E. The population of Camp 1E is 40,000, half of them children under 18 years of age. The average household size is 4 people.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hypertension | 04-06/2020
  Assessment of the prevalence of hypertension in the study groups

SECONDARY OUTCOMES:
Prevalence of diabetes mellitus | 04-06/2020
  Assessment of the prevalence of increased levels of fasting glucose in the study groups
Mean systolic BP | 04-06/2020
  Mean systolic BP among adults aged 18 years and older.
Mean fasting plasma glucose | 04-06/2020
  Mean fasting plasma glucose among adults aged 18 years and older.
Successful BP treatment | 04-06/2020
  The proportion of adults aged ≥ 18 years with hypertension who have a normal BP (systolic BP <140mmHg and a diastolic BP <90mmHg).
Successful diabetes treatment | 04-06/2020
  The proportion of adults aged ≥ 18 years with diabetes or pre-diabetes who have a HbA1c less than 7.0%. HbA1c will only be assessed in a small subgroup of participants (n = 100).
Overweight and obesity | 04-06/2020
  The proportion of adults aged ≥ 18 years being overweight (25 < BMI < 30) and obese (BMI > 30).
WHODAS 2.0 | 04-06/2020
  Health and disability status within the study population as assessed by the WHO Disability Assessment Schedule (WHODAS 2.0).
PHQ-9 | 04-06/2020
  The proportion of adults aged ≥ 18 years with symptoms of depression assessed by the Patient Health Questionnaire (PHQ-9).
CAPS-5 | 04-06/2020
  The proportion of adults aged ≥ 18 years with symptoms of post-traumatic stress disorder assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). CAPS-5 will only be done in a small subgroup of randomly selected participants (n = 100).

CONTACTS AND LOCATIONS:
Overall Officials: Kashem Shaikh, PhD, Principal Investigator — Gono Bishwabidyalay; Alexander Supady, Dr. med. MPH, Principal Investigator — University of Freiburg